CLINICAL TRIAL: NCT00828048
Title: International Registry for Intraductal Papillary Mucinous Neoplasma
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Michele D. Lewis, M.D., PI, Mayo Clinic
Other Study IDs: 07-007845
Record Dates: First submitted 2009-01-21; First posted 2009-01-23 (Estimated); Last update posted 2019-11-06 (Actual); Status verified 2019-11

CONDITIONS: Pancreatic Cysts
MeSH Terms: conditions — Pancreatic Cyst

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pancreatic Cyst: Pancreatic Cyst

SUMMARY:
A centralized web-based database will be used to track patients with IPMN lesions of the pancreas to study natural history and risk factors for malignant transformation in this multi-center study.

DETAILED DESCRIPTION:
Intraductal papillary mucinous neoplasms of the pancreas (IPMN) are increasingly recognized in clinical practice. They represent a unique clinicopathologic entity that is characterized by mucin production, cystic dilation of the pancreatic ducts, and intraductal papillary growth. The World Health Organization recognized IPMN as a distinct clinical entity in 1996. Recent literature suggests that up to 45% of IPMN are malignant and should be resected; however these data are based on larger, primarily symptomatic lesions. Several studies have been published in the recent literature reporting single-center experience with IPMN resections and observations with small numbers of patients. The natural history of these lesions and risk of malignancy is still vague. Consensus guidelines for management of IPMN were published in 2006, but noted the limited knowledge available in six areas: definition and classification, preoperative evaluation, indication for resection, method of resection, histological data on frozen section/positive margins and specimen processing, and finally, method of follow-up. Speaking to this need, we propose an international registry for multi-center collaboration in the above areas of need in IPMN research and clinical management. This will be through a centralized, web-based registry with data entered by each center in a de-identified way to protect confidentiality.

The data collected from the IRB approved retrospective chart review IRB# 07-007202 will be incorporated into this data base. Any patients that participate in the prospective study will be consented with HIPPA consent prior to collection of data.

ELIGIBILITY:
Inclusion Criteria:

* Suspected IPMN based on the consensus guidelines (7)
* Endoscopic ultrasound imaging at baseline examination
* Either surgical histology or clinical follow up with EUS, MRI, or CT scan for at least 1 year
* Cases previously collected that meet the above criteria will be allowed

Exclusion Criteria:

* Patients who do not meet the above inclusion criteria

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary care
Sampling Method: Non-Probability Sample
Enrollment: 290 (Actual)
Dates: Start 2008-03; Primary Completion 2019-11-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
Identify clinical and morphological predictors of cancer or high grade dysplasia in patients with IPMN. Identify predictors of progression to cancer or high grade dysplasia among patients who are followed in surveillance programs. | End of study
  Size and growth pattern of pancreas cysts, presence of mural nodules, development of solid tumor or malignancy will be tracked over time, based on imaging studies including EUS, MRI or CT as clinically indicated.

CONTACTS AND LOCATIONS:
Overall Officials: Michele D Lewis, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Jacksonville, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials